CLINICAL TRIAL: NCT00131521
Title: Comparison of Different Mucoactive Agents for the Care of the Intubated Patient in a Surgical Trauma Intensive Care Unit: A Randomized, Double Blind, Controlled Trial
Brief Title: Comparison of Different Mucoactive Agents for the Care of the Intubated Patient in a Surgical Trauma Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 034-1502-320
Record Dates: First submitted 2005-08-17; First posted 2005-08-18 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Mucus Obstruction; Intubation
Keywords: mucus obstruction, ventilator management
MeSH Terms: interventions — Acetylcysteine; Sodium Chloride

INTERVENTIONS:
Drug: mucomyst
Drug: sodium chloride (saline)

SUMMARY:
This study compares N-acetylcysteine (mucomyst) and sodium chloride to determine their efficacy in the prevention of pulmonary mucus obstruction and retention in intubated patients admitted to the surgical trauma intensive care unit (STICU).

ELIGIBILITY:
Inclusion Criteria:

* Intubated and admitted to the Surgical Trauma Intensive Care Unit (STICU)
* Subjects must be eligible to start treatment within 24 hours of their initial intubation

Exclusion Criteria:

* Patient anticipated to be extubated within 24 hours following STICU admission
* Hypersensitivity to acetylcysteine.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2005-01; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
prevention of pulmonary mucus obstruction

SECONDARY OUTCOMES:
days of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: John G. Myers, M.D., Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Univesity Hospital, San Antonio, Texas, United States